CLINICAL TRIAL: NCT05756998
Title: New Method of IUD Insertion During Cesarian Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: MS-673-2021
Record Dates: First submitted 2023-01-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Contraception
Keywords: IUD; cesarian section; expulsion; postpartum
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic technique (Active Comparator)
  Interventions: Device: Copper T380 IUD ( Paragard 380 A ,CooperSurgical, Inc. © 2022) (classic technique); Procedure: cesarian section
- new technique (Experimental)
  Interventions: Device: Copper T380 IUD ( Paragard 380 A ,CooperSurgical, Inc. © 2022) ( New technique); Procedure: cesarian section

INTERVENTIONS:
Device: Copper T380 IUD ( Paragard 380 A ,CooperSurgical, Inc. © 2022) (classic technique) — During CS , placement of CuT380 IUD at the top of the uterine fundus with ring forceps or manually; before closing the uterine incision, the strings were placed in the lower uterine segment. If the cervix was closed, dilatation from above with ring forceps or manually. Strings passed through the cervix with ring forceps, then checking that IUD remains at the fundus of the uterus prior to closing the uterine incision. The surgeon took a good care not to include IUD strings within the sutures. Six weeks postpartum; Patients will be questioned for any symptoms of complications or side effects. Pelvic examination (per speculum) and transvaginal ultrasound will be performed. Patient satisfaction will be assessed: pain using (VAS score), missed threads.
  Arms: classic technique
Device: Copper T380 IUD ( Paragard 380 A ,CooperSurgical, Inc. © 2022) ( New technique) — During CS, the plunger will be removed, the introducer remains in place and the arms of the IUD were released to be in a transverse position. The introducer will be inserted in the cervical canal through the uterine incision, threads might be shortened if needed or if couldn't be advanced into the cervical canal, The introducer containing the IUD will be then pushed upwards , towards the uterine fundus.The IUD will be placed at the uterine fundus and the IUD will be stabilized at its fundal position by grasping the fundus between the thumb anteriorly and the other fingers posteriorly. The uterine incision was closed while the introducer is in situ , then the introducer will be removed vaginally at the end of CS. Six weeks postpartum; Patients will be followed as in the classic technique group.
  Arms: new technique
Procedure: cesarian section — Under general or spinal anathesia , the abdomen is opened in layers , the bladder is dissected downwards . The uterus is incised at its lower segment & the fetus is extracted , followed by the placenta & membranes . The CU T 380 IUD is inserted either by the classic technique or the standard technique . The uterus is closed in 2 layers by continous non - locked sutures .Proper hemostasis & closure of the abdomen in layers .

SUMMARY:
In women undergoing elective CS, half of them will have Intra-caesarian copper T 380 IUD insertion using the standard method and the remaining half will undergo copper T 380 IUD insertion during CS using a new technique in order to detect which technique is more effective in having more accurate IUD position with visible threads.

DETAILED DESCRIPTION:
Intrauterine device (IUD) is considered one of the most acceptable and effective contraceptive methods used. It is widely accepted and used in Egypt at a large scale than any other type of contraception with many advantages over the other types of contraceptive methods including long acting hormonal methods . Despite IUD complications, it remains the most accepted method, as it has many advantages like being non-coital related, had no systemic complications, of long duration and reversible with rapid return of fertility after its removal . The complications of IUD include heavy menstrual bleedings, menstrual irregularities and infection complications which could be minimized by using strict aseptic techniques during insertion . The most distressing complication is the displacement of IUD, especially if this displacement was extra-uterine, as the patient needs a surgical maneuver (endoscopic usually) for extraction of this IUD. Displacement of IUDs puts a financial and psychological burden to the patient also increases the risk of unwanted pregnancies and its related risks . Displacement of IUD occurs mainly during its insertion, and occurs mainly due to rough or wrong technique; also IUD insertion at a wrong timing may increase risk of IUD displacement. So it is very important to insert IUDs at the proper time with the proper technique . Timing of insertion of IUD after cesarean section is a matter of debate, some gynecologists insert IUDs during cesarean section after placental removal, while other gynecologists prefer insertion of IUDs after an interval either immediately after puerprium (42 days), or after 6 months post-cesarean section, but the majority inserts IUDs after 3 months from cesarean section . The idea of waiting a three-month interval after cesarean section is to assure that the scar had completely healed and the uterus involutes completely to its pre-pregnancy size. The drawbacks of waiting this long interval are poor accessibility of the cervix which may be pulled upward in some cases of repeated cesarean section and loss of self-enthusiasm for rapid contraception after delivery .

ELIGIBILITY:
Inclusion Criteria:

* pregnant , full term patients , scheduled for elective CS.

Exclusion Criteria:

* contraindications for IUD insertion ( chorioamnionitis , congenital uterine malformations ) - Patient refusing IUD contraception.
* Patients with intra-operative bleeding or vital instability.
* Active genital infection at time of insertion.
* Medical disorders e.g. : cardiac , bleeding disorders , T.B. .. etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant patients attending to kasr Alainy Obstetrics and Gynecology Hospital for caesarian section .
Enrollment: 156 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
accuracy of IUD position. | 3 months
  using ultrasound the position of IUD by measuring the distance between the IUD & the fundus of the uterus.
visibility of the threads of IUD. | 3 months
  using a cusco speculum , the IUD threads are inspected.

SECONDARY OUTCOMES:
complications of IUD | 1 month
  complications as pain , vaginal bleeding , infection are followed using specific questionnaire filled by the patient
patient overall satisfaction about the new technique | 3 months
  using specific questionnaire to be filled by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient infertility clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cleland J, Ali M, Benova L, Daniele M. The promotion of intrauterine contraception in low- and middle-income countries: a narrative review. Contraception. 2017 Jun;95(6):519-528. doi: 10.1016/j.contraception.2017.03.009. Epub 2017 Mar 30. PMID 28365165
- [Background] Goldstuck ND, Steyn PS. Insertion of intrauterine devices after cesarean section: a systematic review update. Int J Womens Health. 2017 Apr 18;9:205-212. doi: 10.2147/IJWH.S132391. eCollection 2017. PMID 28458581
- [Background] Sunder, G. and Snigdha, G. (2016) Displaced Intrauterine Device: A Retrospective Study. The Journal of Medical Research, 2, 41-43.